CLINICAL TRIAL: NCT04800458
Title: Contribution of Anti-platelet Antibodies Identified With" Monoclonal Antibody Immobilization of Platelet Antigens" Assay (MAIPA) in the Demonstration of the Auto-immune Character of a Thrombocytopenia at Diagnosis
Brief Title: Contribution of Anti-platelet Antibodies Identified With MAIPA Assay in the Demonstration of the Auto-immune Character of a Thrombocytopenia at Diagnosis
Acronym: APAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/61
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Thrombocytopenia; Immune Thrombocytopenia; Myelodysplasia
Keywords: Monoclonal antibody immobilization of platelet antigens assay; MAIPA; Anti-platelet antibodies; Thrombopoietin
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic; Anemia, Refractory, with Excess of Blasts; Jacobs syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thrombocytopenic patients (Experimental)
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — * Thrombopoietin : 7 ml whole blood.
  * Anti-platelet antibodies free : 14 ml whole blood.
  * Anti-platelet antibodies bound :
  If the platelet count is ≥ 50 G / L : 14 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation ; If the platelet count is < 50 G / L and ≥ 20 G / L : 28 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation ; If the platelet count is < 20 G / L and ≥ 10 G / L: 42 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation ; If the platelet count is < 10 G / L : 49 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation.

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune disease but, paradoxically, and unlike other autoimmune diseases, antiplatelet antibodies are not used either for the diagnosis of the disease or for its prognosis. ITP is a diagnosis of exclusion retained after elimination of other pathologies leading to a thrombocytopenia. No major study has prospectively evaluated the diagnostic value of the presence of anti-platelet antibodies in the etiological investigation of a thrombocytopenia, nor the impact of platelet antibodies on the course of ITP. The gold standard analysis for the determination of platelet antibodies, is the "monoclonal antibody immobilization of platelet antigens" assay (MAIPA), either direct to detect autoantibodies attached to platelets, or indirect to detect circulating antiplatelet antibodies. Therefore, this work aims to study the contribution of the presence of anti-platelet antibodies detected in MAIPA to determine the autoimmune nature of a thrombocytopenia at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old;
* Patients with thrombocytopenia <100 G/L, checked twice, having ruled out false thrombocytopenia by platelet aggregation and acute leukemia by smear;
* No treatment started;
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and prior to any review required by the research);
* Person affiliated or benefiting from a social security scheme.

Exclusion Criteria:

* Secondary ITP;
* False thrombocytopenia;
* Patients who have been transfused with platelets for less than 7 days with efficacy;
* Patient treated for thrombocytopenia (48 hours of corticosteroid therapy is tolerated and is not an exclusion criteria);
* Patient with acute leukemia;
* Pregnant or breastfeeding woman;
* False thrombocytopenia;
* Patient under guardianship, curatorship or any other legal protection regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a diagnosis of autoimmune thrombocytopenia among those in whom will be identified anti-platelet antibodies in direct and indirect MAIPA | 12 months after baseline

SECONDARY OUTCOMES:
Percentage of patients with chronic ITP | 12 months after baseline
serum Thrombopoietin concentration | At baseline and 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François VIALLARD, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de médecine interne, Pessac, France

IPD SHARING:
Plan to Share IPD: No